CLINICAL TRIAL: NCT04238260
Title: Enhancing Physical Therapy Best Practice for Improving Walking After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Janice Eng, Professor, University of British Columbia
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: H19-02809
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Cerebral Infarction; Brain Ischemia; Infarction, Brain
Keywords: Stroke; Lower extremity; Rehabilitation; Wearable device; Exercise; Clinical Trial
MeSH Terms: conditions — Stroke; Cerebral Infarction; Brain Ischemia; Brain Infarction; Motor Activity

STUDY DESIGN:
Intervention Model Description: This clinical trial uses a stepped-wedge design. Unlike typical studies where participants are randomized to two different interventions, this design has all sites start in the Usual Care period, and then switch-over to Enhanced Care at predetermined times, which will then be the new Usual Care (termed "Enhanced Usual Care").
Who Masked: Outcomes Assessor
Masking Description: Assessors at each site will be blinded to intervention. Site study coordinators will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Physical Therapy Care (Active Comparator): Physical Therapists continue usual care
  Interventions: Behavioral: Physical Therapy Usual Care
- Enhanced Physical Therapy Usual Care (Experimental): Best practice implemented
  Interventions: Behavioral: Enhancing Physical Therapy Usual Care

INTERVENTIONS:
Behavioral: Enhancing Physical Therapy Usual Care — The protocol is focused on the completion of a minimum of 30 minutes of weight-bearing, walking-related activities that progressively increase in intensity informed by heart rate and step counters over 4 weeks.
  Arms: Enhanced Physical Therapy Usual Care
Behavioral: Physical Therapy Usual Care — Usual physical therapy
  Arms: Usual Physical Therapy Care

SUMMARY:
The aim of this study is to assess the effect of implementing best practices into current stroke rehabilitation physical therapy on walking outcomes. Participants will also be provided an activity monitor to help them track and target their walking practice to determine if this can improve walking ability.

DETAILED DESCRIPTION:
This multi-site study will have each site start in usual care with participants consented to collecting outcome measures. The twelve inpatient stroke units include: Kelowna General Hospital, Nanaimo Regional General Hospital, Glenrose Rehabilitation Hospital, Saskatoon City Hospital, Wascana Rehabilitation Centre, Joseph Brant Hospital, Bruyère Hospital, Freeport Grand River Hospital, CIUSSS-de-l'Estrie-CHUS Centre de réadaptation de l'Estrie, Centre interdisciplinaire de recherche en réadaptation et intégration sociale, Dr. Everett Chalmers Regional Hospital, and Queen Elizabeth Hospital. Each site will randomly switch over to Enhanced Usual Care (best practice implementation) where all physical therapists at the site will be educated on delivery of best practice for locomotor retraining. The specific therapy activities are at the discretion of the physical therapist; however, physical therapists must work towards thirty minutes of weight-bearing/stepping activity at greater than forty percent heart rate reserve. Participants will continue to be consented to collecting outcome measures. Additionally, participants will be given and trained to use activity watches to monitor their own progress.

ELIGIBILITY:
Inclusion Criteria:

* Admitted by inpatient or day stroke rehabilitation
* Improved walking is a rehabilitation goal
* Within 12 weeks post hemorrhagic or ischemic CVA with hemiparesis (confirmed by medical chart or motor assessment)
* Able to ambulate at least 5 steps. May use assistive and/or orthotic device and maximum one person assist
* Overground walking speed slower than normal
* Able to understand and follow directions
* Greater than or equal to 19 years of age
* Medically stable

Exclusion Criteria:

* Pre-stroke health included a serious gait disorder or disease that affected ambulation (musculoskeletal conditions, amputation, surgery/arthroplasty in the last 6 months, etc.)
* Pre-stroke health included a neurological condition (such as Parkinson's disease or Multiple Sclerosis) or other serious medical condition (active cancer, uncontrolled diabetes)
* Excessive pain in the body/joint preventing participation in an exercise intervention
* Participating in an experimental drug field study
* Participating in another formal exercise rehabilitation clinical trial
* Expected to receive <2 weeks daily in-/out- patient rehabilitation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2021-04-25 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Six-minute walk Test | 4 weeks
  This test measures distance a participant can walk in 6 minutes.

SECONDARY OUTCOMES:
Six-minute walk test | 12 months post-stroke
  This test measures distance a participant can walk in 6 minutes.
Blood pressure | 4 weeks & 12 months post-stroke
  Blood pressure measures physiological effects of the intervention
Euro-QOL 5D-5L | 4 weeks & 12 months post-stroke
  This test is the most widely used instrument to measure quality of life.
Montreal Cognitive Assessment | 4 weeks & 12 months post-stroke
  This test measures levels of cognitive function.
Short performance physical battery | 4 weeks & 12 months post-stroke
  This test measures levels of lower extremity function.
Patient Health Questionnaire-9 (PHQ-9) | 4 weeks & 12 months post-stroke
  This test screens for depression
Modified Rankin Scale (mRS) | 4 weeks & 12 months post-stroke
  This scale measures the degree of disability. Score range: minimum 0 to maximum 6. Lower score means a better outcome.
Physical Activity Scale for the Elderly (PASE) | 12 months post-stroke
  This test assesses physical activity, including leisure, household, and occupational activity. Score range: minimum 0 to maximum 400 or more. Higher score means a better outcome
Step activity monitor | 12 months post stroke
  The number of steps per day over 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Janice J Eng, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
If required by journal for publication, the following individual participant data will be entered into a repository: age in years, sex, and outcomes as described above.

REFERENCES:
- [Derived] Ackerley S, Hung SH, Sheehy L, Donkers SJ, Timofeeva P, Best KL, Peters S, Park SS, Ouellet B, Ezeugwu VE, Milot MH, Sakakibara BM, Eng JJ, Connell LA. Exploring factors influencing implementation across the explanatory-to-pragmatic trial continuum: a sequential qualitative integration of delivering higher-intensity walking exercise within inpatient stroke rehabilitation. Implement Sci Commun. 2026 Jan 8. doi: 10.1186/s43058-025-00812-y. Online ahead of print. PMID 41508158
- [Derived] Hung SH, Ackerley S, Connell LA, Bayley MT, Best KL, Donkers SJ, Dukelow SP, Ezeugwu VE, Milot MH, Peters S, Sakakibara BM, Sheehy L, Yao J, Eng JJ. Real-World Experiences of Therapy Staff Implementing an Intensive Rehabilitation Protocol in Canadian Stroke Inpatient Rehabilitation Settings: A Multi-Site Survey Study. Phys Ther. 2025 Oct 1;105(10):pzaf111. doi: 10.1093/ptj/pzaf111. PMID 41139309
- [Derived] Yan Y, Eng JJ, Hung SH, Bayley MT, Best KL, Connell LA, Donkers SJ, Dukelow SP, Ezeugwu VE, Milot MH, Sakakibara BM, Sheehy L, Wong H, Yao J, Peters S. Aerobic minutes and step number remain low in inpatient stroke rehabilitation. PLoS One. 2025 Jul 28;20(7):e0328930. doi: 10.1371/journal.pone.0328930. eCollection 2025. PMID 40720450
- [Derived] Peters S, Hung SH, Bayley MT, Best KL, Connell LA, Donkers SJ, Dukelow SP, Ezeugwu VE, Milot MH, Sakakibara BM, Sheehy L, Wong H, Yang Y, Yao J, Eng JJ. Safety and effectiveness of the Walk 'n Watch structured, progressive exercise protocol delivered by physical therapists for inpatient stroke rehabilitation in Canada: a phase 3, multisite, pragmatic, stepped-wedge, cluster-randomised controlled trial. Lancet Neurol. 2025 Aug;24(8):643-655. doi: 10.1016/S1474-4422(25)00201-7. PMID 40683274